CLINICAL TRIAL: NCT04728620
Title: A Patient Portal Intervention to Address Diabetes Care Gaps: A Usability Study
Brief Title: Evaluation of a Patient Portal Intervention to Address Diabetes Care Gaps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, William Martinez, MD, MS, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 202281; R18DK123373-01 (NIH)
Record Dates: First submitted 2021-01-21; First posted 2021-01-28 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Medical Informatics; Preventative Care
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will have access to a new feature within an established patient portal native app on mobile devices. The new feature aims to address diabetes care gaps.
  Interventions: Other: Diabetes Care Gaps Patient Portal Intervention

INTERVENTIONS:
Other: Diabetes Care Gaps Patient Portal Intervention — The Diabetes Care Gaps Patient Portal Intervention involves a new feature embedded with the My Health At Vanderbilt (MHAV) native app (on Epic's MyChart platform) for mobile devices that allows patients to: (a) receive notifications when the patient is due for certain types of diabetes monitoring and preventative care and (b) initiate an order for the care. Automated notifications will be sent to patients if, according to the evidence-based guidelines, the patients are due for a hemoglobin A1C blood test, microalbumin urine test, diabetes eye exam, or pneumonia vaccination. Once notified patients can initiate orders for the care within the MHAV app. The patient will receive confirmation when the order has been processed and will be provided instructions to receive the relevant care.

SUMMARY:
The purpose of this study is to evaluate the usability of a novel patient portal intervention designed to: (a) notify patients when selected, clinically meaningful, evidence-based diabetes monitoring & preventative care (e.g., annual diabetes eye exam) become due and (b) allow patients to initiate orders for the care. In addition, the investigators will assess pre-post change on secondary psychosocial outcomes (e.g., self-efficacy).

DETAILED DESCRIPTION:
Up to 60 adult patients with type 1 or 2 diabetes mellitus will be enrolled and given access to a new feature within the patient portal at Vanderbilt University Medical Center. The new feature will be available via the patient portal native app (i.e., My Health at Vanderbilt (MHAV) app) for mobile devices (smartphone or tablet). The new feature will allow patients to: (1) receive notifications when the patient is due for certain types of diabetes monitoring and preventative care and (2) initiate an order for the care.

Study participants will complete questionnaires electronically via email at three time points: baseline (T0), immediately after first use of the intervention (T1), and three-month follow-up (T2) to as assess study outcomes including usability and pre-post change in secondary psychosocial outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Established patient at participating primary care clinic
* Type 1 or 2 diabetes mellitus
* Able to speak and read in English
* Age 18 to 75 years old
* Mobile device (smartphone or tablet) with internet access
* Active MHAV account and willing and able to use the MHAV native app on a mobile device
* Due (based on evidence-based guidelines) for any of the following: hemoglobin A1C, urine microalbumin, diabetes eye exam, and/or pneumococcal vaccination.

Exclusion Criteria:

* Known cognitive deficits or functional impairment preventing the use of a mobile device
* Pregnant or planning to become pregnant during the study period
* Severe difficulty seeing
* Severe difficulty hearing
* Medical condition that make it hard for people to understand what they are saying

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Martinez, MD, MS, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
After study results are posted on clinical trials and published in a peer-reviewed journal, de-identified individual participant data that underlie the results reported will be available upon requests made to the principal investigator and ending after 36 months after publication.
Supporting Information: Study Protocol, SAP
Time Frame: Deidentified individual participant data that underlie the results reported will be available after publication in a peer reviewed journal and posted on clinical trials and ending after 36 months after publication.
Access Criteria: Researchers should provide a methodologically sound proposal to achieve their proposed aims. Proposals may be submitted to the principal investigator up to 36 months following publication. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 60 enrolled participants, 50 completed the baseline questionnaire and still had at least one diabetes care gap (due for any of the following: hemoglobin A1C, urine microalbumin, diabetes eye exam, and/or pneumococcal vaccination) and were then assigned to the intervention.
Period: Overall Study
Arm/Group | Intervention
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 30
  Black or African American | 15
  Other | 5
Region of Enrollment [Number; unit: participants]
  United States | 50
Health Literacy [Count of Participants; unit: Participants]
  Adequate Health Literacy | 36
  Limited Health Literacy | 14

OUTCOME MEASURES:

1. Primary Outcome: Usability
Description: The System Usability Scale (SUS) is a validated measure of usability. The ten items are scored on a five-point Likert scale. The item scores are summed and then converted to a score ranging from 0 (worst) to 100 (best). A score of above 68 indicative of "above average" usability.
Time Frame: Immediately after first use T(1), at approximately 1 month
Population: 36 participants used to the study intervention during the study period and completed the SUS scale after first use.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 36
score on a scale | 79.3 (14.9)
Statistical Analysis 1: Comparison: Intervention; One-sample t-test comparing the sample mean to the threshold value of 71 indicative of "good" usability. The null hypothesis: true mean is 71 or less; Test type: Superiority — single group; p = 0.001, t-test, 1 sided; mean = 79.3

2. Primary Outcome: User Experience
Description: User experience will be assessed by study-specific survey items administered to all participants at the end of the study period (T2). The survey items will inquire about participants' perspectives on the acceptability of the intervention and on particular components of the intervention such as notifications.
Time Frame: 3-month follow up (T2)
Population: Not all patients completed this item on the final questionnaire (T2), results limited to the 47 who responded to the items.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 47
Participants
  Would recommend the intervention to other patients: Strongly agree/agree | 37
  Would recommend the intervention to other patients: Neutral/disagree/strongly disagree | 10
  Would continue to use the intervention in future if it remained available: Strongly agree/agree | 38
  Would continue to use the intervention in future if it remained available: Neutral/disagree/strongly disagree | 9

3. Secondary Outcome: Change in Attitudes Toward Managing Diabetes in General
Description: The 5-item Manage Disease in General Scale of the Chronic Disease Self-Efficacy Scales is a validated measure of self-efficacy (i.e., the confidence a person has in managing their own health and health care) and is closely related to patient activation. The items were adapted to be specific to diabetes rather than a generic condition or illness. Each item uses a 10-point Likert-type scale of response options ranging from 1 (not at all confident) to 10 (totally confident). The score for the scale is the mean of the items. Higher scores indicate greater self-efficacy.
Time Frame: Enrollment (T0) and 3-month follow up (T2)
Population: 4 participants did not complete the Manage Disease in General Scale on the three-month follow-up post-questionnaire and were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 46
score on a scale
  baseline questionnaire (T0) | 8.1 (1.5)
  three-month follow-up questionnaire (T2) | 8.6 (1.2)
Statistical Analysis 1: Comparison: Intervention; Test type: Other; p = 0.005, t-test, 2 sided; Mean Difference (Net) = 0.57

4. Secondary Outcome: Change in Diabetes Distress
Description: The Problem Areas in Diabetes Scale (PAID-5) is a valid measure of diabetes distress. Total scores on the PAID-5 can range from 0 to 20, with higher scores suggesting greater diabetes-related emotional distress.
Time Frame: Enrollment (T0) and 3-month follow up (T2)
Population: 4 participants did not complete the Problem Areas in Diabetes Scale (PAID-5) on the three-month follow-up post-questionnaire and were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 46
score on a scale
  baseline questionnaire (T0) | 6.6 (5.0)
  three-month follow-up questionnaire (T2) | 5.8 (4.9)
Statistical Analysis 1: Comparison: Intervention; Test type: Other; p = 0.19, t-test, 2 sided; Mean Difference (Net) = -0.85

5. Secondary Outcome: Change in Understanding of Diabetes Monitoring and Preventative Care
Description: Unique study specific items to assess participants' understanding of measures of diabetes monitoring and preventative care (e.g., Diabetes Eye Exams) will be administered to all study participants.
Time Frame: Enrollment (T0) and 3-month follow up (T2)
Population: Not all patients answers all Understanding of Diabetes Monitoring and Preventative Care items on both the baseline (T0) and three-months (T2). Participants with missing this data at either time point were excluded from the analysis with up to 5 participants missing data for one of items.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 46
Participants
  Correctly identify the recommended frequency of A1c monitoring at baseline (T0) | 38
  Correctly identify the recommended frequency of A1c monitoring at three-months (T2) | 38
  Correctly identify the recommended frequency of urine microalbumin screening at baseline (T0) | 24
  Correctly identify the recommended frequency of urine microalbumin screening at three-months (T2) | 23
  Correctly identify the recommended frequency of pneumonia vaccination at baseline (T0): number analyzed (Participants) | 45
  Correctly identify the recommended frequency of pneumonia vaccination at baseline (T0) | 13
  Correctly identify the recommended frequency of pneumonia vaccination at three-months (T2): number analyzed (Participants) | 45
  Correctly identify the recommended frequency of pneumonia vaccination at three-months (T2) | 13
  Correctly identify the recommended frequency of diabetes eye exams at baseline (T0) | 45
  Correctly identify the recommended frequency of diabetes eye exams at three-months (T2) | 45
Statistical Analysis 1: Comparison: Intervention; Analysis for pre-post change in knowledge of recommended A1c monitoring frequency; Test type: Other; p = 1, McNemar
Statistical Analysis 2: Comparison: Intervention; Analysis for pre-post change in knowledge of recommended urine microalbumin screening frequency; Test type: Other; p = 1, McNemar
Statistical Analysis 3: Comparison: Intervention; Analysis for pre-post change in knowledge of recommended pneumonia vaccination frequency; Test type: Other; p = 1, McNemar
Statistical Analysis 4: Comparison: Intervention; Analysis for pre-post change in knowledge of recommended diabetes eye exam frequency; Test type: Other; p = 1, McNemar

6. Secondary Outcome: Patient Initiated Orders
Description: The investigators will collect data on the number of patient-initiated orders for evidence-based diabetes monitoring and preventative services (e.g., hemoglobin A1c). Participants with more than one diabetes care gap can initiated an order for more than one evidence-based diabetes monitoring and preventative service (e.g. hemoglobin A1c and diabetes eye exam).
Time Frame: 3-month follow up (T2)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 50
Participants
  Initiated order for hemoglobin A1c | 14
  Initiated order for urine microalbumin | 17
  Initiated order for pneumococcal vaccination | 6
  Initiated order for diabetes eye exam | 10

7. Secondary Outcome: Order Completion
Description: The investigators will collect data on the number of completed (i.e., care received) evidence-based diabetes monitoring and preventative services after a corresponding patient initiated order.
Time Frame: 3-month follow up (T2)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 50
Participants
  Completed a hemoglobin A1c lab test after patient initiated order | 13
  Completed a urine microalbumin lab test after patient initiated order | 15
  Completed a pneumococcal vaccination after patient initiated order | 6
  Completed a diabetes eye exam after patient initiated order | 5

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 3/50
Other Adverse Events (participants affected / at risk) | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=50)
Hospitalization (General disorders) | 3 (5) — Not related to study participation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/20/NCT04728620/Prot_SAP_001.pdf
  • Informed Consent Form (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT04728620/ICF_000.pdf